CLINICAL TRIAL: NCT00922103
Title: A Historical Cohort Study, to Investigate Morbidity, Functional and Physiological Outcome, as Well as Endoscopic and Histological Aspects and the Quality of Life, of the Ileo Neo Rectal Anastomosis (INRA) Compared to the Ileo Pouch Anal Anastomosis (IPAA), for Patients With Ulcerative Colitis (UC)
Brief Title: A Study to Investigate the Ileo Neo Rectal Anastomosis Compared to the Ileo Pouch Anal Anastomosis for Patients With Ulcerative Colitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elisabeth-TweeSteden Ziekenhuis (Other)
Collaborators: Radboud University Medical Center (Other)
Responsible Party: JT Heikens, MD, St Elisabeth Hospital, Tilburg, The Netherlands
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0426; AMO nr. 04/074
Record Dates: First submitted 2009-06-12; First posted 2009-06-17 (Estimated); Last update posted 2010-09-13 (Estimated); Status verified 2010-09

CONDITIONS: Colitis, Ulcerative; Surgery
Keywords: Colitis, Ulcerative; Ileo Neo Rectal Anastomosis; Ileal Pouch Anal Anastomosis; Quality of Life; functional results; reconstructive surgery; surgery
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Proctocolectomy, Restorative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- INRA (Experimental): Patients treated for medical refractory Ulcerative Colitis
  Interventions: Procedure: Ileal Neo Rectal Anastomosis
- IPAA (Active Comparator): Patients treated for medical refractory Ulcerative Colitis
  Interventions: Procedure: Ileal Pouch Anal Anastomosis

INTERVENTIONS:
Procedure: Ileal Neo Rectal Anastomosis — Comparison of the Ileal Neo Rectal Anastomosis to the Ileal Pouch Anal Anastomosis in patients treated for medical refractory Ulcerative Colitis
  Arms: INRA
Procedure: Ileal Pouch Anal Anastomosis — Comparison of the Ileal Pouch Anal Anastomosis to the Ileal Neo Rectal Anastomosis in patients treated for medical refractory Ulcerative Colitis
  Arms: IPAA

SUMMARY:
For patients with ulcerative colitis, eligible for surgical treatment, which restorative surgical procedure: the standard ileo pouch anal anastomosis or the alternative ileo neo rectal anastomosis is the best in terms of complications, functional outcome and health status and quality of life.

DETAILED DESCRIPTION:
This research is designed to answer questions from the medical profession and patients´ community (Crohn en Colitis Ulcerosa Society, the Netherlands) whether the new INRA technique needs further development on a broader scale or not.

The research project will be conducted in the two institutes where INRA procedures have been carried out and in the UMCN to recruit matched control IPAA patients. There is a large experience with the IPAA procedure in this latter institute. The University of Tilburg will participate to work on health status and quality of life aspects. They have a large experience with quality of life research in general and have participated in QOL research in this topic before.

The aim of this historical cohort study is to establish the value of INRA, compared to IPAA, for patients with ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

* UC patients with INRA procedure
* Age, sex and disease specific matched group of UC-IPAA patients with temporary diverting ileostomy from the same period
* Written informed consent

Exclusion criteria

* Pregnancy
* Malignancy (apart from basalioma or carcinoma-in-situ of cervix)
* Psychiatric disease or inability to assess follow up

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2005-06; Primary Completion 2009-12 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
functional outcome | after surgery: 3 months, 6 months, 12 months and yearly afterwards
Quality of life and Health Status | after surgery: 3 months, 6 months, 12 months and yearly afterwards

SECONDARY OUTCOMES:
histo-pathologic results | after surgery: 3 months, 6 months, 12 months and yearly afterwards
endoscopic results | after surgery: 3 months, 6 months, 12 months and yearly afterwards
morbidity and mortality | after surgery: 3 months, 6 months, 12 months and yearly afterwards
ano-rectal physiology | after surgery: 3 months, 6 months, 12 months and yearly afterwards

CONTACTS AND LOCATIONS:
Overall Officials: JT Heikens, MD, Principal Investigator — St Elisabeth Hospital, Tilburg, The Netherlands; D de Jong, MD, PhD, Study Chair — University Medical Centre St Radboud, Nijmegen, The Netherlands; JLJM Teepen, MD, PhD, Study Chair — St Elisabeth Hospital, Tilburg, The Netherlands; JHJM van Krieken, MD, PhD, Study Chair — University Medical Centre St Radboud, The Netherlands; HG Gooszen, MD, PhD, Study Chair — University Medical Centre St Radboud, Nijmegen, The Netherlands; J de Vries, Md, PhD, Study Chair — St Elisabeth Hospital, Tilburg, The Netherlands; CJHM van Laarhoven, MD, PhD, Study Director — University Medical Centre St Radboud, The Netherlands
Locations (2):
- Netherlands (2):
  - University Medical Centre St Radboud, Nijmegen, Gelderland
  - St Elisabeth Hospital, Tilburg, North Brabant